CLINICAL TRIAL: NCT01734512
Title: PNOC 001: Phase II Study of Everolimus for Recurrent or Progressive Low-grade Gliomas in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Pacific Pediatric Neuro-Oncology Consortium (Other); The Pediatric Low Grade Astrocytoma (PLGA) Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120817; NCI-2012-02774 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Recurrent Progressive Low-grade Gliomas; Pediatric Progressive Low-grade Gliomas
Keywords: pediatric recurrent progressive low-grade gliomas; pediatric progressive low-grade gliomas; everolimus; mTOR inhibition
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Everolimus (Experimental): Everolimus tablet will be taken daily by mouth with water. Twenty-eight days will constitute one course and subsequent courses will immediately follow with no break in the administration of the drug. Dosing is based on the body surface area (BSA) calculated at the beginning of each course of therapy. Patients will also be provided with a drug diary for everolimus. The maximum time on study is 24-months, but if there is no disease progression or adverse events, the patient may speak with a doctor about continuing the treatment off-study.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus tablet will be taken daily by mouth with water. All participants will be given a dose of 5 mg/m2/dose daily.
  Other Names: Zortress; Afinitor

SUMMARY:
This is an open label study of everolimus in children with recurrent or progressive low-grade glioma.

DETAILED DESCRIPTION:
This is an open label study of everolimus in children with recurrent or progressive low-grade glioma. All patients will receive everolimus at a dose of 5 mg/m2/dose daily. An adaptive Simon two-stage design for phase 2 studies of targeted therapies will be used to assess the efficacy primary objective. The proposed treatment with everolimus will be deemed not worthy of further investigation in this patient population if the true PFS at 6-months (PFS6) is less than 50%. If in the first stage, with a combined sample size of 25, there is preliminary evidence to suggest efficacy of everolimus is restricted to patients with PI3K/AKT/mTOR activation as measured by p-S6 positivity, a total of 45 patients will be enrolled and the design will have 81% statistical power to detect a true disease stabilization rate ≥70%. If in the first stage there is preliminary evidence to suggest efficacy of everolimus is independent of PI3K/AKT/mTOR activation, a total of 65 patients will be enrolled and the design will have >95% statistical power to detect a true disease stabilization rate ≥70%.

ELIGIBILITY:
Inclusion Criteria:

--Patients must have radiographic progressive or recurrent confirmed world health organization (WHO) grade I or II astrocytomas, that was confirmed histologically. Progressive or recurrent disease should be based on MRI according to the definition below.

Eligible histologies:

* Pilocytic Astrocytoma - 90600112
* Astrocytoma, Low Grade (Fibrillary astrocytoma, WHO Grade 2) - 10065886
* Astrocytoma, Low Grade (Low-grade Astrocytoma, not otherwise specified (NOS), WHO Grade 2) - 10003571

  * Tissue from the initial diagnosis or recurrence must be made available for correlative testing.
  * Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least two dimensions on MRI.
  * Patients may have had treatment (chemotherapy and/or radiotherapy) for any number of relapses prior to this recurrence.
  * Patients must have received their last dose of myelosuppressive anticancer chemotherapy at least three (3) weeks prior to study registration or at least six (6)weeks of nitrosourea.
  * Patients must have received their last dose of other investigational or biological agent > 7 days prior to study entry.

For agents that have known adverse events occurring beyond 7 days after administration, this period should be extended beyond the time during which adverse events are known to occur. This should be discussed with the study chair.

* If patients received prior monoclonal antibody treatment, at least three half-lives must be elapsed by the time of treatment initiation. These patients should also be discussed with the study chair.
* Patients must have received their last fraction of craniospinal or focal radiation to primary tumor or other sites >12 weeks (3 months) prior to registration.

  --Age ≥3 and ≤21 years.
* Because no dosing or adverse event data are currently available on the use of everolimus in patients <3 years of age, these young children are excluded from this study.

  * Life expectancy of greater than 8 weeks.
  * Patients must be able to swallow pills.
  * Patient must have a Karnofsky (if ≥ 16 years of age) or Lansky Performance score (if ≤ 16 years of age) of ≥50 by the time of registration.
  * Patients must have adequate bone marrow function (ANC ≥ 1,000/mm3, platelet count of ≥ 100,000/mm3, and hemoglobin ≥ 9 gm/dL) before starting therapy. Eligibility level for hemoglobin may be reached by transfusion.
  * International Normalized Ratio (INR) ≤1.5. (Anticoagulation is allowed if target INR ≤ 1.5 on a stable dose of warfarin or on a stable dose of low molecular weight (LMW) heparin for >2 weeks at time of randomization).
  * Patients must have adequate liver function (SGPT/alanine aminotransferase (ALT) ≤ 2.5 times ULN and bilirubin ≤ 1.5 times ULN) before starting therapy.
  * Patients must have adequate renal function (serum creatinine ≤ 1.5 times institutional ULN for age or Glomerular filtration rate (GFR) ≥ 70 ml/min/1.73 m2) before starting therapy.
  * Patients must have cholesterol level <350 mg/dL and triglycerides < 400 mg/dL before starting therapy. In case one or both of these are exceeded, the patient can only be included after initiation of appropriate lipid lowering medication and documentation of cholesterol < 350mg/dL and triglycerides < 400mg/dl before start of therapy.
  * Patients must have normal pulmonary function testing for age based on pulse oximetry.
  * The effects of everolimus on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because everolimus are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
  * Female patients of child bearing potential must not be breastfeeding or pregnant as evidenced by a negative pregnancy test.

Exclusion Criteria:

* Patients with primary spinal cord tumors
* Patients receiving concomitant medication that may interfere with study outcome. For example, patients cannot be on enzyme inducing anticonvulsants like phenytoin.
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, bacille Calmette-Guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* Hepatitis B/C blood test must be done at screening for all patients. Patients who test positive for Hepatitis C antibodies and the Hepatitis B antigen are ineligible.
* A known history of HIV seropositivity. HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with everolimus. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Patients receiving chronic, systemic treatment with corticosteroids or another immunosuppressive agent. Topical or inhaled corticosteroids are allowed.
* Patients may not have therapy for this recurrence (including radiation).
* Patients who do not have measurable disease on MRI.
* Patients who have been previously treated with an mTOR inhibitor.
* Patients with a known hypersensitivity to everolimus or other rapamycins (e.g. sirolimus, temsirolimus).
* Patients receiving any other concurrent anticancer or investigational therapy.
* Patients with any clinically significant unrelated systemic illness that would compromise the patient's ability to tolerate protocol therapy.
* Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection.
* Patients with inability to return for follow-up visits to assess toxicity to therapy.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years.

Note: A detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients. Hepatitis B Virus (HBV) DNA and Hepatitis C Virus (HCV) RNA Polymerase chain reaction (PCR) testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV/HCV infection.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2012-12-13 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2024-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Haas-Kogan, MD, Study Chair — Dana-Farber Cancer Institute; Sabine Mueller, MD, Principal Investigator — University of California, San Francisco
Locations (18):
- United States (18):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - Children's Hospital Oakland, Oakland, California
  - University of California, San Diego Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Children's Hospitals and Clinics of Minneapolis, Minneapolis, Minnesota
  - St. Louis Children's Hospital, Washington University, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - The Children's Hospital Of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - University of Utah, Salt Lake City, Utah
  - University of Washington, Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haas-Kogan DA, Aboian MS, Minturn JE, Leary SES, Abdelbaki MS, Goldman S, Elster JD, Kraya A, Lueder MR, Ramakrishnan D, von Reppert M, Liu KX, Rokita JL, Resnick AC, Solomon DA, Phillips JJ, Prados M, Molinaro AM, Waszak SM, Mueller S. Everolimus for Children With Recurrent or Progressive Low-Grade Glioma: Results From the Phase II PNOC001 Trial. J Clin Oncol. 2024 Feb 1;42(4):441-451. doi: 10.1200/JCO.23.01838. Epub 2023 Nov 17. PMID 37978951

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus: Everolimus tablet will be taken daily by mouth with water. Twenty-eight days will constitute one course and subsequent courses will immediately follow with no break in the administration of the drug. Dosing is based on the body surface area (BSA) calculated at the beginning of each course of therapy. Patients will also be provided with a drug diary for everolimus. The maximum time on study is 24-months, but if there is no disease progression or adverse events, the patient may speak with a doctor about continuing the treatment off-study.
  Everolimus: Everolimus tablet will be taken daily by mouth with water. All patients will be given a dose of 5 mg/m2/dose daily.
Period: Overall Study
Arm/Group | Everolimus
Started | 65
Completed | 65
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 65
Age, Customized [Count of Participants; unit: Participants]
  3-9 years old | 35
  10-21 years old | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 47
  More than one race | 1
  Unknown or Not Reported | 14
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression Free Survival at 6 Months
Description: Response was be determined by bi-dimensional diameters. RECIST criteria will be collected and used for secondary evaluation. Patients will have brain MRI scans with and without gadolinium performed prior to therapy, after every second course in the first year, after every third course in the second year, and at the End of Study visit (if not done within prior 3 months). Spine MRIs should be performed prior to therapy and at the same time points as standard brain MRIs if clinically indicated.
Time Frame: Up to 6 months
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Everolimus
Number analyzed (Participants) | 65
percentage | 67 [54 to 77]

2. Secondary Outcome: Proportion of Participants With Objective Response
Description: The proportion of participants who demonstrated a complete or partial response as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1 Criteria where Complete Response (CR) is defined as the complete disappearance of all known disease for >=8 weeks. Complete response is dated from time all lesions have disappeared on a stable or decreasing dose of corticosteroids. A Partial Response (PR) is a reduction of at least 50% in the size of all measurable tumor as quantitated by sum of the products of the largest diameters (SLD) of measurable lesions and maintained for >=8 weeks on a stable or decreasing dose of corticosteroids. Partial response is dated from the time of first observation. Overall response also takes into account the response in both the target and non-target lesion, and the appearance of new lesions, where applicable and depend on the achievement of both measurement and confirmation criteria.
Time Frame: Up to 6 months
Measure: Number; unit: proportion of participants
Arm/Group | Everolimus
Number analyzed (Participants) | 65
proportion of participants | 0.05

3. Secondary Outcome: Median Progression Free Survival in Recurrent Pediatric Low-grade Glioma (LGGs)
Description: Progression free survival will be calculated from date of first treatment to the date of first observation of progressive disease, non-reversible neurological progression or increasing steroid requirements (applies to stable disease only), death due to any cause, or early discontinuation of treatment
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Everolimus
Number analyzed (Participants) | 65
days | 365 [225 to 765]

4. Secondary Outcome: Median Overall Survival From Time of Diagnosis
Description: Overall survival in participants with recurrent pediatric low-grade glioma (LGGs) will be calculated from date of original diagnoses to death using Kaplan Meier method. Median time to death and 95% confidence interval will be reported.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Everolimus
Number analyzed (Participants) | 65
days | NA [NA to NA] — Less than 50% of the participants died at the time study data collection ended, so a median survival time could not be calculated due to the insufficient number of events.

5. Secondary Outcome: Median Overall Survival From Time of Enrollment
Description: Overall survival in participants with recurrent pediatric low-grade glioma (LGGs) will be calculated from date of study registration to death using Kaplan Meier method. Median time to death and 95% confidence interval will be reported.
Time Frame: Up to 5 years
Population: Less than 50% of the participants died at the time study data collection ended, so a median survival time could not be calculated due to the insufficient number of events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Everolimus
Number analyzed (Participants) | 65
days | NA [NA to NA] — Less than 50% of the participants died at the time study data collection ended, so a median survival time could not be calculated as the curve did not drop below the level of detection.

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Everolimus
All-Cause Mortality (participants affected / at risk) | 9/65
Serious Adverse Events (participants affected / at risk) | 20/65
Other Adverse Events (participants affected / at risk) | 62/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=65)
Edema face (General disorders) | 1 (1)
Hearing Impaired (Ear and labyrinth disorders) | 1 (1)
Seizure (Nervous system disorders) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hydrocephalus (Nervous system disorders) | 6 (12)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Skin infection (Skin and subcutaneous tissue disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (5)
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 2 (5)
Hypertension (Vascular disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=65)
Cholesterol high (Investigations) | 34 (63)
Aspartate aminotransferase increased (Investigations) | 30 (62)
Alanine aminotransferase increased (Investigations) | 26 (60)
Neutrophil count decreased (Investigations) | 19 (41)
Lymphocyte count decreased (Investigations) | 15 (25)
White blood cell decreased (Investigations) | 15 (49)
Platelet count decreased (Investigations) | 14 (23)
Investigations - Other (Investigations) | 11 (27)
Weight loss (Investigations) | 6 (8)
Alkaline phosphatase increased (Investigations) | 6 (7)
Creatinine increased (Investigations) | 4 (8)
Mucositis oral (Gastrointestinal disorders) | 35 (94)
Diarrhea (Gastrointestinal disorders) | 15 (30)
Nausea (Gastrointestinal disorders) | 14 (16)
Vomiting (Gastrointestinal disorders) | 11 (12)
Oral pain (Gastrointestinal disorders) | 8 (11)
Abdominal pain (Gastrointestinal disorders) | 7 (8)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 (6)
Stomach pain (Gastrointestinal disorders) | 4 (7)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 34 (98)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (30)
Hypophosphatemia (Metabolism and nutrition disorders) | 15 (23)
Hypokalemia (Metabolism and nutrition disorders) | 13 (35)
Anorexia (Metabolism and nutrition disorders) | 9 (12)
Hypernatremia (Metabolism and nutrition disorders) | 9 (18)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 6 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (7)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (11)
Headache (Nervous system disorders) | 21 (35)
Dizziness (Nervous system disorders) | 5 (5)
Fatigue (General disorders) | 25 (36)
Fever (General disorders) | 10 (19)
Pain (General disorders) | 4 (4)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (17)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 5 (5)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (9)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Anemia (Blood and lymphatic system disorders) | 18 (47)
Upper respiratory infection (Infections and infestations) | 8 (9)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 4 (5)
Sinus tachycardia (Cardiac disorders) | 8 (17)
Hypertension (Vascular disorders) | 6 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT01734512/Prot_SAP_000.pdf